CLINICAL TRIAL: NCT04813887
Title: Skin Diseases: Which Heathcare Professionals do Pregnant Women in Vendee Use?
Brief Title: Skin Diseases and Pregnancy: Which Heathcare Professionals ?
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD21_0020
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-03

CONDITIONS: Skin Abnormalities; Pregnancy
MeSH Terms: conditions — Skin Abnormalities | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Self-questionnaire on skin diseases reported during pregnancy

SUMMARY:
Pregnancy-induced physiological dermatological changes are common. In 2016, they represented between 23% (acne) and 75% (pigmentary changes) of pregnancies in France. Some dermatological changes require medical advice to identify a possible pathological rash.

These pathological rashes can be dangerous for the mother or the fetus.

The aim of this study is to assess the prevalence of skin diseases during pregnancy and to evaluate the care pathway in a healthcare sector (Vendee) for these pregnant women?

DETAILED DESCRIPTION:
Pregnancy-induced physiological dermatological changes are common. In 2016, they represented between 23% (acne) and 75% (pigmentary changes) of pregnancies in France. Some dermatological changes require medical advice to identify a possible pathological rash.

These pathological rashes can be dangerous for the mother or the fetus. It is therefore essential to recognize them for a quick specialized treatment. They include: intrahepatic cholestasis of pregnancy, pemphigoid gestationis, polymorphic eruption during pregnancy, atopic eczema, generalized pustular psoriasis in pregnancy.

In view of the demography of dermatologists in the Vendee, 18 dermatologists in 2020 in all establishments (hospitals, clinics, practices), the general practitioner is at the center of these considerations.

The aim of this study is to assess the situation of skin disease during pregnancy and to evaluate the care pathway in a healthcare sector (Vendee) for these pregnant women?

ELIGIBILITY:
Inclusion Criteria:

* Any woman who gives birth at Departmental Hospital Center of Vendee

Exclusion Criteria:

* Patient's refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective collection of data from a questionnaire answered by patients giving birth at the Departmental Hospital Center of Vendee during the postpartum period.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Identify the health care provider that pregnant women consult when experiencing a skin disease | after delivery during the patient's stay in the maternity (2-3 days)
  Type of health care provider seeing a pregnant woman for skin disease

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, Principal Investigator — Departmental Hospital Center of Vendee
Locations (1):
- CHD Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No